CLINICAL TRIAL: NCT06776679
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-BGB-16673 Following a Single Oral Dose in Healthy Male Participants
Brief Title: A Study of How [14C]-BGB-16673 is Absorbed, Broken Down, and Removed From the Body After a Single Oral Dose in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-16673-106
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm: [14C]-BGB-16673 (Experimental): Participants will receive a single dose of [14C]-BGB-16673
  Interventions: Drug: [14C]-BGB-16673

INTERVENTIONS:
Drug: [14C]-BGB-16673 — Administered orally as suspension in lipid vehicle

SUMMARY:
The purpose of this study is to determine the absorption, metabolism, and excretion of [14C]-BGB-16673 and to characterize and determine, where possible, the metabolites present in plasma, urine, and feces in healthy male participants following a single oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m², inclusive.
* Good health, as determined by no clinically significant findings from medical history.
* History of a minimum of 1 bowel movement per day.
* Able to comprehend and are willing to sign the Informed Consent Form (ICF) and abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* Confirmed systolic blood pressure >140 or <90 mmHg, diastolic blood pressure >90 or <50 mmHg, or pulse rate >100 or <40 beats per minute.
* Alcohol consumption of >21 units per week for males.
* Positive urine drug screen at screening or positive alcohol test result or positive urine drug screen at check-in.
* Ingestion of caffeine-containing foods or beverages within 48 hours of check-in or intend to ingest caffeine-containing foods or beverages until end of study.
* Use of tobacco- or nicotine-containing products within 3 months prior to check-in, or positive cotinine at screening or check-in.
* Ingestion of Seville orange- or grapefruit-containing foods or beverages within 7 days prior to check-in.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Total Radioactivity Recovery (fet1-t2) in Urine and Feces | Approximately 35 Days
Area Under the Plasma Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC0-∞) of BGB-16673 | Approximately 35 Days
Area Under the Plasma Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC0-∞) for Total Radioactivity in Plasma and Whole Blood | Approximately 35 Days
Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast) of BGB-16673 | Approximately 35 Days
Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast) for Total Radioactivity in Plasma and Whole Blood | Approximately 35 Days
Maximum Observed Plasma Concentration (Cmax) of BGB-16673 | Approximately 35 Days
Maximum Observed Plasma Concentration (Cmax) for Total Radioactivity in Plasma and Whole Blood | Approximately 35 Days
Time of the Maximum Observed Plasma Concentration (Tmax) of BGB-16673 | Approximately 35 Days
Time of the Maximum Observed Plasma Concentration (Tmax) for Total Radioactivity in Plasma and Whole Blood | Approximately 35 Days
Apparent Terminal Elimination Half-life (t1/2) of BGB-16673 | Approximately 35 Days
Apparent Terminal Elimination Half-life (t1/2) for Total Radioactivity in Plasma and Whole Blood | Approximately 35 Days
Urinary recovery of BGB-16673 (fet1-t2) | Approximately 35 Days
Quantitative metabolic profiles of BGB-16673 in plasma and excreta | Approximately 35 Days
Identification of BGB-16673 major metabolites in plasma and excreta | Approximately 35 Days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Approximately 35 days
Number of Participants with Clinically Significant Laboratory Values | Approximately 9 weeks
Number of Participants with Clinically Significant Electrocardiogram (ECG) Results | Approximately 9 weeks
Number of Participants with Clinically Significant Vital Sign Measurements | Approximately 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Study Director, Study Director — BeiGene
Locations (1):
- Fortrea Clinical Research Unit Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/